CLINICAL TRIAL: NCT05058105
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single- and Multiple Ascending-dose Study of the Safety, Tolerability, and Pharmacokinetics of Intravenous FL058 and Meropenem Alone and in Combination in Healthy Chinese Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics of Intravenous FL058 and Meropenem in Healthy Subjects(SAD/MAD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FL058-I-03
Record Dates: First submitted 2021-09-08; First posted 2021-09-27 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Healthy
MeSH Terms: interventions — Meropenem

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- FL058 500mg and Meropenem 1000mg (Experimental): FL058 500mg and Meropenem 1000mg (8 subjects);
  FL058 Placebo and Meropenem 1000mg(2 subjects)
  Interventions: Drug: FL058 500mg and Meropenem 1000mg（ IV 120min）; Drug: FL058 Placebo and Meropenem 1000mg（ IV 120min）
- FL058 1000mg and Meropenem 1000mg (Experimental): D1
  FL058 1000mg(8 subjects) and FL058 Placebo(2 subjects);
  D4
  Meropenem 1000mg(8 subjects) and Meropenem Placebo(2 subjects);
  D7~ D15
  FL058 1000mg and Meropenem 1000mg (8 subjects);
  FL058 Placebo and Meropenem 1000mg(2 subjects)
  Interventions: Drug: FL058 1000mg（ IV 120min）; Drug: FL058 Placebo （ IV 120min）; Drug: Meropenem 1000 mg （ IV 120min）; Drug: Meropenem Placebo （ IV 120min）; Drug: FL058 1000mg and Meropenem 1000mg （ IV 120min）; Drug: FL058 Placebo and Meropenem 1000mg （ IV 120min）
- FL058 1000mg and Meropenem 2000mg (IV 120min) (Experimental): FL058 1000mg and Meropenem 2000mg (8 subjects);
  FL058 Placebo and Meropenem 2000mg(2 subjects)
  Interventions: Drug: FL058 1000mg and Meropenem 2000mg （ IV 120min）; Drug: FL058 Placebo and Meropenem 2000m（ IV 120min）
- FL058 1000mg and Meropenem 2000mg (IV 180min) (Experimental): FL058 1000mg and Meropenem 2000mg (8 subjects);
  FL058 Placebo and Meropenem 2000mg(2 subjects)
  Interventions: Drug: FL058 1000mg and Meropenem 2000mg （ IV 180min）; Drug: FL058 Placebo and Meropenem 2000m（ IV 180min）
- FL058 2000mg and Meropenem 2000mg (Experimental): FL058 2000mg and Meropenem 2000mg (8 subjects);
  FL058 Placebo and Meropenem 2000mg(2 subjects)
  Interventions: Drug: FL058 2000mg and Meropenem 2000mg（ IV 180min）; Drug: FL058 Placebo and Meropenem 2000mg（ IV 180min）

INTERVENTIONS:
Drug: FL058 500mg and Meropenem 1000mg（ IV 120min） — D1 qd;
  D2~ D8 q8h;
  D9 qd
  Arms: FL058 500mg and Meropenem 1000mg
Drug: FL058 Placebo and Meropenem 1000mg（ IV 120min） — D1 qd;
  D2~ D8 q8h;
  D9 qd
  Arms: FL058 500mg and Meropenem 1000mg
Drug: FL058 1000mg（ IV 120min） — D1 qd;
  Arms: FL058 1000mg and Meropenem 1000mg
Drug: FL058 Placebo （ IV 120min） — D1 qd;
  Arms: FL058 1000mg and Meropenem 1000mg
Drug: Meropenem 1000 mg （ IV 120min） — D4 qd;
  Arms: FL058 1000mg and Meropenem 1000mg
Drug: Meropenem Placebo （ IV 120min） — D4 qd;
  Arms: FL058 1000mg and Meropenem 1000mg
Drug: FL058 1000mg and Meropenem 1000mg （ IV 120min） — D7 qd;
  D8~ D14 q8h;
  D15 qd;
  Arms: FL058 1000mg and Meropenem 1000mg
Drug: FL058 Placebo and Meropenem 1000mg （ IV 120min） — D7 qd;
  D8~ D14 q8h;
  D15 qd;
  Arms: FL058 1000mg and Meropenem 1000mg
Drug: FL058 1000mg and Meropenem 2000mg （ IV 120min） — D1 qd;
  D2~ D8 q8h;
  D9 qd
  Arms: FL058 1000mg and Meropenem 2000mg (IV 120min)
Drug: FL058 Placebo and Meropenem 2000m（ IV 120min） — D1 qd;
  D2~ D8 q8h;
  D9 qd
  Arms: FL058 1000mg and Meropenem 2000mg (IV 120min)
Drug: FL058 1000mg and Meropenem 2000mg （ IV 180min） — D1 qd;
  D2~ D8 q8h;
  D9 qd
  Arms: FL058 1000mg and Meropenem 2000mg (IV 180min)
Drug: FL058 Placebo and Meropenem 2000m（ IV 180min） — D1 qd;
  D2~ D8 q8h;
  D9 qd
  Arms: FL058 1000mg and Meropenem 2000mg (IV 180min)
Drug: FL058 2000mg and Meropenem 2000mg（ IV 180min） — D1 qd;
  D2~ D8 q8h;
  D9 qd
  Arms: FL058 2000mg and Meropenem 2000mg
Drug: FL058 Placebo and Meropenem 2000mg（ IV 180min） — D1 qd;
  D2~ D8 q8h;
  D9 qd
  Arms: FL058 2000mg and Meropenem 2000mg

SUMMARY:
Phase 1 Study of the Safety, Tolerability, and Pharmacokinetics of FL058 and Meropenem Alone and in Combination following Single and Multiple Doses in Healthy Adult Subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged between 18 and 45 years (inclusive).
2. Body mass index (BMI) ranges from 19 to 26 kg/m2 (inclusive), and the body weight is ≥50kg.
3. Good general health as determined by the Investigator based on medical history, physical examination, vital signs, 12-lead ECG and clinical laboratory tests.
4. Provide voluntary written informed consent prior to any study procedures and are willing and able to comply with the prescribed treatment protocol and evaluations.

Exclusion Criteria:

1. Concurrent or history of clinically significant cardiovascular, hepatic, renal, endocrine, gastrointestinal, respiratory, psychiatric, neurologic and/or hematological disorders.
2. Positive screen result for HBsAg, HCV-Ab, or HIV-Ab at screening.
3. History of clinically significant food or drug allergy.
4. A QT interval corrected using Fridericia's formula >450 msec.
5. eGFR<90mL/min/1.73m2.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events [Safety and Tolerability] | Day 1 to Day 24

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital affiliated to Fudan University, Shanghai, China

REFERENCES:
- [Derived] Huang Z, Yang X, Jin Y, Yu J, Cao G, Wang J, Hu Y, Dai J, Wu J, Wei Q, Tian Y, Yu S, Zhu X, Mao X, Liu W, Liang H, Zheng S, Ju Y, Wang Z, Zhang J, Wu X. First-in-human study to evaluate the safety, tolerability, and population pharmacokinetic/pharmacodynamic target attainment analysis of FL058 alone and in combination with meropenem in healthy subjects. Antimicrob Agents Chemother. 2024 Jan 10;68(1):e0133023. doi: 10.1128/aac.01330-23. Epub 2023 Dec 6. PMID 38054726